CLINICAL TRIAL: NCT03240510
Title: Understanding Male Breast Cancer: Salah Azaïz Cancer Institute Experience
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Salah Azaïz Cancer Institute (Other)
Responsible Party: Principal Investigator, Syrine Abdeljaoued, PhD in Oncology, Study Chair, Salah Azaïz Cancer Institute
Other Study IDs: SalahSCI
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Male Breast Cancer
Keywords: Breast cancer; Male
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The goal of this study is to evaluate the Salah Azaïz Cancer Institute male breast cancer patients population over a period of 14 years.

Goal of the retrospective part: to gather clinicopathologic data and follow-up outcomes of male breast cancer patients diagnosed and/or treated at Salah Azaïz Cancer Institute from 2004 to 2013.

Goal of the prospective part: to create a registry of male patients with breast cancer for a period of 48 months (from 2014 to 2017).

ELIGIBILITY:
Inclusion Criteria:

Histological diagnosis of male breast cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective part: All men with histologically proven invasive breast carcinoma diagnosed between 2004 and 2013.
  Prospective part: All men with histologically proven invasive breast carcinoma diagnosed between 2014 and 2017.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes | Through study completion, an average of 4 year
  Survival, Disease free survival
Clinico-biological characteristics of the disease | Through study completion, an average of 4 year

CONTACTS AND LOCATIONS:
Overall Officials: Syrine Abdeljaoued, PhD, Study Chair — Salah Azaïz Cancer Institute; Ilhem Bettaieb, Dr, Principal Investigator — Salah Azaïz Cancer Institute; Amor Gamoudi, Pr, Principal Investigator — Salah Azaïz Cancer Institute
Locations (1):
- Salah Azaïz Cancer Institute, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided